CLINICAL TRIAL: NCT05087394
Title: Cohort of COVID19 Patients Admitted to Pasteur Clinic 2020-2021
Brief Title: COVID19 Hospitilized in Clinica Pasteur of Neuquen (Argentina)
Acronym: COVIDPas
Status: Completed | Type: Observational
Sponsor: Asociacion Latinoamericana de Torax (Industry)
Responsible Party: Principal Investigator, Gustavo Zabert, MD, Principal investigator, Asociacion Latinoamericana de Torax
Other Study IDs: COVIDPas1
Record Dates: First submitted 2021-10-18; First posted 2021-10-21 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Comorbidity; Respiration, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Comorbidities — Risk factors (comorbidities), requirements of respiratory suppot and chest imaging will are considered exposure for primary outcomes
  Other Names: Oxigen requirement; Mechanical Ventilation; High flow nasal cannula; Chest CT scan; CT pulmonary angiogram (CTPA)

SUMMARY:
retrospective cohort (non-experimental study) of COVID 19 patients assisted in hospitalization (severe and critical) between 2020 and 2021

DETAILED DESCRIPTION:
Consecutive patients with acute infection by SARS-COV2 and severe or critical COVID19 disease, or acute complications, hospitalized in the Pasteur Clinic of Neuquén city from the beginning of the pandemic in the region until December 31, 2021. Data were obtained retrospectively from information registered simultaneously with hospitalization in three databases (RedCap, DataTech and Excel).

. Inclusion criteria

* Adult patients (over 18 years old)
* Suffering from acute infection by SARS-Cov2, diagnosed by PCR-real time, detection of viral antigen, specific antibodies with or clinical epidemiological criteria
* Hospitalized defined by attending physicians or referral (severe or critical according to NIH) Exclusion criteria
* Patients under 18 years of age.
* Convalescent from acute SARS-Cov2 infection and without evidence of a new event of reinfection.
* Outpatient management or hospitalization less than 24 hours for diagnosis and / or evaluation of severity or complications. Sample Selection Method First patient was registered at the beginning of the pandemic in the region March 20, 2020) and is expected to recruit the las patient diagnosed in December 31, 2021.

The recruitment is consecutive without other selection criteria.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (over 18 years old)
* Suffering from acute infection by SARS-Cov2, diagnosed by PCR-real time, detection of viral antigen, specific antibodies with or clinical epidemiological criteria
* Hospitalization defined by attending or referral physician (severe or critical according to NIH)

Exclusion Criteria:

* Patients under 18 years of age.
* Convalescent from acute SARS-Cov2 infection and without evidence of a new event reinfection.
* Outpatient management or hospitalization less than 24 hours for diagnosis and / or evaluation of severity or complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with severe or critical (according to NIH) COVID19 diseased admitted to Pasteur Clinic in 202 and 2021
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
28-day mortality | From date of admition until the date of death from any cause, assessed up to 28 day
  defined as death ocurred within 28 days of admition to hospital
Hospital mortality | From date of admition until the date of death from any cause, assessed up to 52 weeks
  defined as death ocurred within hospitalization

SECONDARY OUTCOMES:
Invasive Mechanical ventilation | From date of admition until the date of equirement of invasive mechanical ventilation, assessed up to 21 day
  defined as requirement of invasive mechanical ventilation support

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Zabert, MD, Principal Investigator — Clinica Pasteur; Ignacio Zabert, MD, Study Director — Clinica Pasteur; Ignacio Veltri, MD, Study Director — Clinica Pasteur
Locations (1):
- Pasteur Clinic, Neuquén, Nqn, Argentina

IPD SHARING:
Plan to Share IPD: Undecided
at the end of the study or at specific requirements

REFERENCES:
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Grasselli G, Pesenti A, Cecconi M. Critical Care Utilization for the COVID-19 Outbreak in Lombardy, Italy: Early Experience and Forecast During an Emergency Response. JAMA. 2020 Apr 28;323(16):1545-1546. doi: 10.1001/jama.2020.4031. No abstract available. PMID 32167538
- [Background] Working group for the surveillance and control of COVID-19 in Spain; Members of the Working group for the surveillance and control of COVID-19 in Spain. The first wave of the COVID-19 pandemic in Spain: characterisation of cases and risk factors for severe outcomes, as at 27 April 2020. Euro Surveill. 2020 Dec;25(50):2001431. doi: 10.2807/1560-7917.ES.2020.25.50.2001431. PMID 33334400
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Aylward L, Liang W, Dong X, et al., World Health Organization W. Report of the WHO-China Joint Mission on Coronavirus Disease 2019 (COVID-19). WHO-China Jt Mission Coronavirus Dis 2019. 2020;1(16-24 February):1-40.
- [Background] Lamfre L, Caro P, Hasdeu S, Horne F. Modelo de Proyección de Casos Esperados COVID-19 En Argentina 2020. Neuquen https://1331c255-c873-472c-8edd- 6738111a6c38.filesusr.com/ugd/d623b6_007bc0ad0898495882e61367e1d2644d.pdf.
- [Background] Espinosa L, Ambort C, Vera M, et al. Documento de Comité Asesor de Ética de La Clínica Pasteur Para La Implementación Del Documento de Aspectos Éticos En La Pandemia de COVID19 En El Escenario de Recursos Escasos. Neuquen; 2020. https://drive.google.com/drive/u/0/folders/1BK1rSlpCR2KzydRxRp6KKUsqLezIKsAi
- [Background] MSal Neuquen. ASPECTOS ÉTICOS EN LA ATENCIÓN DE LAS PERSONAS DURANTE LA PANDEMIA POR CORONAVIRUS ( SARS-CoV-2 ). Neuquen; 2020.
- See also: Documento de Comité Asesor de Ética de La Clínica Pasteur Para La Implementación Del Documento de Aspectos Éticos En La Pandemia de COVID19 En El Escenario de Recursos Escasos. Neuquen; 2020 — https://drive.google.com/drive/u/0/folders/1BK1rSlpCR2KzydRxRp6KKUsqLezIKsAi